CLINICAL TRIAL: NCT07326631
Title: Finerenone for Cardiorenal Protection in Diabetic CKD: Impact on Renal Function Decline and Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Muhammad Awais Danish, Dr, Nishtar Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22126
Record Dates: First submitted 2025-12-09; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Kidney Disease (DKD); Heart Failure
MeSH Terms: conditions — Diabetic Nephropathies; Heart Failure | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Finerenone Group (Experimental): Finerenone Drug
  Interventions: Drug: Finerenone

INTERVENTIONS:
Drug: Finerenone — To assess the effect of Finerinone on slowing renal function decline and improving cardiovascular outcomes, particularly heart failure risk, in patients with diabetic CKD.

SUMMARY:
To assess the effect of Finerinone on slowing renal function decline and improving cardiovascular outcomes, particularly heart failure risk, in patients with diabetic CKD.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Diagnosed cases of type 2 diabetes mellitus.
* Chronic kidney disease with eGFR 25-90 mL/min/1.73m² and/or UACR ≥30 mg/g.
* On stable ACE inhibitor or ARB therapy for at least 4 weeks.
* Serum potassium ≤4.8 mmol/L.
* Provided written informed consent.

Exclusion Criteria:

* Symptomatic heart failure (NYHA class II-IV).
* eGFR <25 mL/min/1.73m² or on maintenance dialysis.
* Known non-diabetic kidney disease.
* Recent major cardiovascular event (within 30 days).
* Serum potassium >4.8 mmol/L or history of severe hyperkalaemia.
* Contraindication or hypersensitivity to finerenone.
* Pregnancy or lactation.
* Any condition limiting compliance or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Renal Function Decline post finerinone therapy | From enrollment to the end of treatment at 06 months
  Progressive worsening of kidney function is defined as a sustained ≥40% reduction in eGFR from baseline, progression to kidney failure (ESKD), or renal death.
Number of Participants with Heart Failure (HF) Event post finerinone therapy | 6 month
  Defined as hospitalization for new or worsening heart failure, confirmed by clinical evidence of fluid overload, raised BNP levels and the requirement for intravenous therapy or hemodynamic support.
eGFR Measurement | 06 months
  Estimated glomerular filtration rate calculated using the CKD-EPI formula, standardized for body surface area (mL/min/1.73 m²).
Number of Participants with Albuminuria | 06 months
  Measured as urinary albumin-to-creatinine ratio (UACR), with categories of moderately increased (30-300 mg/g) and severely increased (>300 mg/g) albuminuria, per KDIGO classification used in the trial protocols.
Number of Participants with Hyperkalaemia post treatment | 06 months
  Defined as a serum potassium level >5.5 mmol/L, which served as a safety threshold for dose adjustment or discontinuation in the parent trial data.
Number of Participants with Cardiovascular (CV) Event post treatment with finerinone therapy | 06 months
  Includes CV death, non-fatal myocardial infarction, non-fatal stroke, or hospitalization for heart failure (HHF) - forming the composite cardiovascular outcome measure in the finerenone studies.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.frontiersin.org/journals/cardiovascular-medicine/articles/10.3389/fcvm.2024.1476029/full

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-12-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT07326631/Prot_SAP_ICF_000.pdf